CLINICAL TRIAL: NCT04062513
Title: Effectiveness of Olfactive Stimulation Interventions With Mothers' Milk on Preterm Pain Response: a Randomized Controlled Trial
Brief Title: Olfactive Stimulation Interventions With Mothers' Milk on Preterm Pain Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, De Clifford-Faugère Gwenaelle, Principal investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-21-2020-2309
Record Dates: First submitted 2019-08-12; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Pain, Acute; Preterm Infant; Breast Milk
MeSH Terms: conditions — Acute Pain; Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Olfactive stimulation intervention with familiarization (Experimental): Participants will receive the olfactive stimulation intervention with mothers' milk odor during a previous period of nine hours and during heel prick. Sucrose will be also administered during heel prick.
  Interventions: Other: Olfactive stimulation intervention with familiarization
- Olfactive stimulation intervention (Experimental): Participants will receive the olfactive stimulation intervention with mothers' milk odor during heel prick only. Sucrose will be also administered during heel prick.
  Interventions: Other: Olfactive stimulation intervention
- Standard care (Other): In the control arm, participants will receive the standard care for pain which is sucrose administration.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Olfactive stimulation intervention with familiarization — The intervention consists of placing a pad immersed with breast milk near the preterm infant's nose during heel prick. For the familiarization stage, infants were familiarized with the odor of their mothers' milk for 9 hours before heel prick.
  Arms: Olfactive stimulation intervention with familiarization
Other: Olfactive stimulation intervention — The intervention consists of placing a pad immersed with breast milk near the preterm infant's nose during heel prick.
  Arms: Olfactive stimulation intervention
Other: Standard care — Preterm infants will receive sucrose during heel prick.
  Arms: Standard care

SUMMARY:
Repeated and untreated pain can lead to long-term consequences in preterm infants, such as pain hypersensitivity and impaired motor and intellectual development. Studies on the pharmacological and non-pharmacological interventions for pain management in preterm infants are limited. Thus, we investigated an intervention based on olfactive stimulation with mothers' milk. The aims of this study are: a) Evaluate the effectiveness of an olfactive stimulation intervention with mothers' milk odor on preterm procedural pain; b) Evaluate the effectiveness of adding a period of familiarization previous to the olfactive stimulation intervention with mothers' milk odor on preterm procedural pain. Preterm infants will be recruited and randomly assigned to three groups 1) mothers' milk odor during the nine hours before and during heel-prick, 2) mothers' milk odor during heel-prick, 3) standard care. Pain will be measured using a scale of pain adapted for preterm infants. This procedure with mothers'milk odor is inexpensive and easily performed.This study will significantly contribute to the advancement of knowledge on preterm infants pain management.

ELIGIBILITY:
Inclusion Criteria for mothers

* 18 years or older,
* speak, understand and write French or English
* express their milk

Exclusion Criteria for mothers

- pathology or condition that contraindicates the use of their breast milk (HIV, drugs...)

Inclusion Criteria for preterm

* 29 to 36 weeks of gestation
* APGAR > 6 at 5 minutes
* less than 21 days

Exclusion Criteria for preterm

* intubated, under Continuous Positive Airway Pressure or nasal oxygen,
* surgery in the first day of life
* congenital disease
* intraventricular hemorrhage > grade II
* leukomalacia
* sedation within 48 hours prior to heel prick
* pharmacologic treatment for pain within 12 hours prior to heel prick
* being under phototherapy treatment during the familiarization stage

Ages: 29 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pain : Premature Infant Pain Profile-Revised | Change from baseline every 30 seconds until 120 seconds post heel lance and 30 seconds after the end of blood collection
  Scores range from 0 to 21 where a higher score means more pain, a score less than 6 signifies an absence of pain, and a score greater than 12 indicates moderate to severe pain. The PIPP-R contains four parts: gestational age, state of sleep-awake, physiological parameters, and behavioural parameters.

SECONDARY OUTCOMES:
Recovery | The time required for the preterm infant to return to baseline heart rate levels (should not exceed 5 minutes)
Maternal acceptability of the olfactive stimulation intervention : questionnaire | Immediately post-procedure
  After the intervention, mothers will be asked to complete a questionnaire focusing on maternal acceptability of the olfactive stimulation intervention with mothers' milk to manage procedural pain (demographic questions and Likert scale).

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Aita, PhD, Study Director — Université de Montréal

REFERENCES:
- [Background] De Clifford-Faugere G, Lavallee A, Aita M. Olfactive stimulation interventions for managing procedural pain in preterm and full-term neonates: a systematic review protocol. Syst Rev. 2017 Oct 17;6(1):203. doi: 10.1186/s13643-017-0589-1. PMID 29041964
- [Background] De Clifford-Faugère G, Aita M, Héon M, Le May S. Management of procedural pain in preterm infants through olfactive stimulation with mothers' milk: A pilot study. Science of Nursing and Health Practices - Science infirmière et pratiques en santé. 2(1), Article 3, 2019. Available at: https://doi.org/10.31770/2561-7516.1042